CLINICAL TRIAL: NCT04222894
Title: Hospital Workplace Nutrition Study (Sibley Memorial Hospital)
Brief Title: Hospital Workplace Nutrition Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: Sibley Memorial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00038823
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Overweight; Type2 Diabetes
Keywords: body weight; blood pressure; lipids; nutrition
MeSH Terms: conditions — Overweight; Body Weight | interventions — Diet, Plant-Based; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-based diet (Active Comparator): The diet group will be asked to follow a low-fat, vegan diet for 12 weeks
  Interventions: Other: Plant-based diet
- Control diet (Active Comparator): Half of the participants will be asked to continue their usual diets for the 12-week study period.
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: Plant-based diet — Weekly instructions will be given to the participants in the intervention group about following vegan diet.
  Other Names: Vegan diet
  Arms: Plant-based diet
Other: Control Diet — Participants will be asked to continue their usual diets for the 12-week study period.
  Arms: Control diet

SUMMARY:
The purpose of this study is to evaluate the effects of a plant-based diet on body weight, blood pressure, and plasma lipid concentrations, as part of a hospital workplace program.

DETAILED DESCRIPTION:
Using a randomized controlled trial design, participants will be randomly assigned to either a plant-based or a control diet for 12 weeks. T Before and after each intervention period, the investigators will measure participant body weight, blood pressure, and plasma lipid concentrations.

ELIGIBILITY:
Inclusion Criteria:

1. Employee of Sibley hospital
2. Male or female
3. Age at least 18 years
4. Have a BMI >25 kg/m2
5. Ability and willingness to participate in all components of the study
6. A willingness to follow a plant-based diet for the duration of the study
7. A willingness to attend weekly classes for the duration of the study
8. A willingness to keep physical activity level consistent throughout the duration of the study

Exclusion Criteria:

1. Diabetes mellitus type 1 or history of any endocrine condition that would affect body weight, such as a pituitary abnormality or Cushing's syndrome
2. Smoking during the past six months
3. Alcohol consumption of more than 2 drinks per day or the equivalent, episodic increased drinking (e.g., more than 2 drinks per day on weekends), or a history of alcohol abuse or dependency followed by any current use
4. Current or unresolved past drug abuse
5. Pregnancy or plans to become pregnant in the next 12 weeks
6. Intention to leave hospital employment in the next 12 weeks
7. Unstable medical or psychiatric status
8. Evidence of an eating disorder
9. Lack of English fluency
10. Inability to maintain current medication regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Body Weight | 12 weeks
  Anticipated weight-loss for intervention group compared with control group
Blood Pressure | 12 weeks
  Anticipated changes in blood pressure (systolic and diastolic) for intervention group compared with control group
Plasma Lipids | 12 weeks
  Anticipated changes in plasma lipid concentrations for intervention group compared with control group

SECONDARY OUTCOMES:
Hemoglobin A1c | 12 weeks
  HbA1c will be measured as an index of glycemic control.
Fasting Plasma Glucose | 12 weeks
  Fasting Plasma Glucose will be measured as an index of glycemic control.
Absenteeism | 12 weeks
  Absenteeism from work will be assessed by self-report at baseline and final assessments.
Quality of Life: SF-36 | 12 weeks
  Quality of life will be assessed using the SF-36, which is a brief health survey with 36 questions. The SF-36 provides an 8-scale profile of functional health and well-being scores, as well as psychometrically-based physical and mental health summary measures. The SF-36 is a general measure that has been administered across various age groups, disease spectra, and treatment regimens. Items on the SF-36 are scored on a scale of 0-100, with a higher score indicating better health-related quality of life.
Dietary Restraint, Disinhibition, Hunger | 12 weeks
  Participants will complete an Eating Inventory form, a highly reliable 51 item questionnaire providing quantitative measures of dietary restraint (21 questions), disinhibition (16 items), and hunger (14 questions). Scores for each sub-scale are calculated by summing respective items. The scale consists of 36 true=false items and 15 forced-choice format questions. Higher scores are indicative of greater dietary restraint, disinhibition and hunger. Its principal use in the current study will be as a gauge of ease in adapting to the intervention diet, which is indicated by changes in restraint and hunger scores.
Food Acceptability: The Food Acceptability Questionnaire | 12 weeks
  The Food Acceptability Questionnaire will measure attitudes about the intervention diet, including desire to adhere, likelihood to adhere in the future, and attitudes about accessibility of sustaining the diet. Items on the FAQ are scored on a scale of 1-7. Higher scores indicate greater food acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Neal D Barnard, MD, Principal Investigator — President
Locations (1):
- Sibley Memorial Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Luckhaupt SE, Cohen MA, Li J, Calvert GM. Prevalence of obesity among U.S. workers and associations with occupational factors. Am J Prev Med. 2014 Mar;46(3):237-48. doi: 10.1016/j.amepre.2013.11.002. PMID 24512862
- [Background] Dayoub E, Jena AB. Chronic Disease Prevalence and Healthy Lifestyle Behaviors Among US Health Care Professionals. Mayo Clin Proc. 2015 Dec;90(12):1659-62. doi: 10.1016/j.mayocp.2015.08.002. Epub 2015 Oct 5. PMID 26422242
- [Background] Vibhute NA, Baad R, Belgaumi U, Kadashetti V, Bommanavar S, Kamate W. Dietary habits amongst medical students: An institution-based study. J Family Med Prim Care. 2018 Nov-Dec;7(6):1464-1466. doi: 10.4103/jfmpc.jfmpc_154_18. PMID 30613543
- [Background] Bergeron N, Al-Saiegh S, Ip EJ. An Analysis of California Pharmacy and Medical Students' Dietary and Lifestyle Practices. Am J Pharm Educ. 2017 Oct;81(8):5956. doi: 10.5688/ajpe5956. PMID 29200450
- [Background] Bleich SN, Bennett WL, Gudzune KA, Cooper LA. Impact of physician BMI on obesity care and beliefs. Obesity (Silver Spring). 2012 May;20(5):999-1005. doi: 10.1038/oby.2011.402. Epub 2012 Jan 19. PMID 22262162
- [Background] Barnard ND, Scialli AR, Bertron P, Hurlock D, Edmonds K, Talev L. Effectiveness of a low-fat vegetarian diet in altering serum lipids in healthy premenopausal women. Am J Cardiol. 2000 Apr 15;85(8):969-72. doi: 10.1016/s0002-9149(99)00911-x. PMID 10760336
- [Background] Yokoyama Y, Nishimura K, Barnard ND, Takegami M, Watanabe M, Sekikawa A, Okamura T, Miyamoto Y. Vegetarian diets and blood pressure: a meta-analysis. JAMA Intern Med. 2014 Apr;174(4):577-87. doi: 10.1001/jamainternmed.2013.14547. PMID 24566947
- [Background] Barnard ND, Cohen J, Jenkins DJ, Turner-McGrievy G, Gloede L, Jaster B, Seidl K, Green AA, Talpers S. A low-fat vegan diet improves glycemic control and cardiovascular risk factors in a randomized clinical trial in individuals with type 2 diabetes. Diabetes Care. 2006 Aug;29(8):1777-83. doi: 10.2337/dc06-0606. PMID 16873779
- [Background] Esselstyn CB Jr. Updating a 12-year experience with arrest and reversal therapy for coronary heart disease (an overdue requiem for palliative cardiology). Am J Cardiol. 1999 Aug 1;84(3):339-41, A8. doi: 10.1016/s0002-9149(99)00290-8. PMID 10496449
- [Background] Esselstyn CB Jr, Ellis SG, Medendorp SV, Crowe TD. A strategy to arrest and reverse coronary artery disease: a 5-year longitudinal study of a single physician's practice. J Fam Pract. 1995 Dec;41(6):560-8. PMID 7500065
- [Background] Ornish D, Brown SE, Scherwitz LW, Billings JH, Armstrong WT, Ports TA, McLanahan SM, Kirkeeide RL, Brand RJ, Gould KL. Can lifestyle changes reverse coronary heart disease? The Lifestyle Heart Trial. Lancet. 1990 Jul 21;336(8708):129-33. doi: 10.1016/0140-6736(90)91656-u. PMID 1973470
- [Background] Craig WJ, Mangels AR; American Dietetic Association. Position of the American Dietetic Association: vegetarian diets. J Am Diet Assoc. 2009 Jul;109(7):1266-82. doi: 10.1016/j.jada.2009.05.027. PMID 19562864
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Loffler A, Luck T, Then FS, Sikorski C, Kovacs P, Bottcher Y, Breitfeld J, Tonjes A, Horstmann A, Loffler M, Engel C, Thiery J, Villringer A, Stumvoll M, Riedel-Heller SG. Eating Behaviour in the General Population: An Analysis of the Factor Structure of the German Version of the Three-Factor-Eating-Questionnaire (TFEQ) and Its Association with the Body Mass Index. PLoS One. 2015 Jul 31;10(7):e0133977. doi: 10.1371/journal.pone.0133977. eCollection 2015. PMID 26230264